CLINICAL TRIAL: NCT02293772
Title: Planetary Habitat Simulation: An Investigation Into the Effects of Hypoxia and / or Bedrest on Fuel Metabolism and Appetite (WP5)
Brief Title: Planetary Habitat Simulation: Nutrition Studies
Acronym: PlanHab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Jozef Stefan Institute (Other); KTH Royal Institute of Technology (Other); European Commission (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 284438/WP5
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Hypoxia
Keywords: Bedrest; Appetite
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypoxic ambulatory (Active Comparator): Ambulatory in normobaric hypoxia
  Interventions: Other: Hypoxic ambulatory
- Hypoxic Bedrest (Experimental): Bedrest in normobaric hypoxia
  Interventions: Other: Hypoxic Bedrest
- Normoxic bedrest (Active Comparator): Bedrest in normobaric normoxia
  Interventions: Other: Normoxic Bedrest

INTERVENTIONS:
Other: Hypoxic ambulatory — 21 days confinement in normobaric hypoxic (FiO2 = 14%) environment
  Arms: Hypoxic ambulatory
Other: Hypoxic Bedrest — 21 days supine bedrest in normobaric hypoxic (FiO2 = 14%) environment
  Arms: Hypoxic Bedrest
Other: Normoxic Bedrest — 21 days supine bedrest in normobaric normoxic (FiO2 = 21%) environment
  Arms: Normoxic bedrest

SUMMARY:
A loss of body weight has been documented in lowland-living individuals when exposed to hypoxic environments, such as at high altitude, or under laboratory conditions. A reduction in appetite and energy intake has also been reported during conditions of microgravity, such as during space flight. Fourteen normal or over-weight men, who are otherwise healthy, will undergo 3x 21-day interventions; normobaric normoxic bed rest (NBR; FiO2=21%), normobaric hypoxic ambulatory confinement (HAMB; FiO2=14%; ~4000 m simulated altitude), and normobaric hypoxic bed rest (HBR; FiO2=14%). The effects of hypoxia and bedrest on appetite and its hormonal control will be assessed before and at day 17 of each intervention using a mixed meal tolerance test.

DETAILED DESCRIPTION:
A loss of body weight has been documented in lowland-living individuals when exposed to hypoxic environments, such as at high altitudes, or under laboratory conditions. This weight loss has been attributed both to a reduced appetite (and subsequent fall in dietary energy intake), and to an increase in resting energy expenditure. Interestingly, a reduction in appetite and energy intake has also been reported during space flight, although the mechanism for this has not been explained. As the gas inside future planetary habitats is likely to have lower partial pressure of oxygen than in Earth's atmospheric air, hypoxia induced appetite reduction could pose a challenge for individuals in these environments. For example, persistent under-eating could compromise long term health due to inadequate intake of essential micronutrients, especially in the presence of altered nutrient metabolism and requirements seen during space flight. Moreover, inadequate macronutrient intake could exacerbate the loss of lean body tissue which occurs in situations (such as microgravity, inactivity and bed rest) where muscles are unloaded. Indeed, a protein intake greater than normal could be required in situations where there is muscle inactivity, to achieve the same postprandial anabolic effect of amino acids seen in ambulatory individuals.

The mechanism for the reduction in appetite observed in hypoxia is not well established. Several incretin hormones and adipokines have been implicated in the control of appetite and may be candidates for inducing this alteration in appetite observed in hypoxia. However, reports in the literature present contradictory findings, perhaps due to the use of different experimental paradigms (hypobaric and normobaric hypoxia, active and resting subjects, variability in the degree and duration of hypoxia).

The protocol of the current study standardises physical activity, ambient temperature, hypoxic stimulus and nutritional composition of the diet, and aims to extend our knowledge of the effects of hypoxia and bedrest on appetite and its hormonal control.

In order to discern the separate and combined effects of microgravity and hypoxia, fourteen normal or over-weight men, who are otherwise healthy, will be recruited following medical and psychological screening. They will be invited to attend the Olympic Sport Centre, Planica, Slovenia on 3 occasions, with each visit being 31 days in duration and separated by 5 months. Each 31-day visit ('campaign') includes a baseline recording period (5 days), 21 days of intervention and a recovery period (5 days), with the 3 interventions allocated in a randomized, cross over design: i) Normobaric normoxic bed rest (NBR; FiO2=21%), ii) Normobaric hypoxic ambulatory confinement (HAMB; FiO2=14%; ~4000 m simulated altitude), and iii) Normobaric hypoxic bed rest (HBR; FiO2=14%). A standardized, repeating, 14-day dietary menu, comprised of foods commonly consumed in the Slovenian diet, will be applied during all campaigns, the targeted energy intakes being calculated individually using a modified Benedict-Harris formula with physical activity factor multipliers of 1.2 for the HBR and NBR campaigns and 1.4 for the HAMB campaign. Food will be provided in weighed portions and subjects will be encouraged to eat all food supplied. However, any food not eaten will be weighed and actual amount consumed recorded in a diet analysis programme. Body mass will be assessed daily during the campaigns using a gurney incorporating load cells, and whole body composition will be determined before and immediately after each intervention using fan beam dual-emission X-ray absorptiometry.

Participants will undergo a mixed meal tolerance test before and on day 17 of each intervention period, in the morning, after a 12 hour fast, with the time of assessment replicated on each study day at every campaign. On arrival, participants will rest supine on a hospital bed and place their hand in a heated hand warming unit (air temperature 50-55oC). An intravenous cannula will then be inserted retrograde into a dorsal hand vein for arterialised-venous blood sampling. After 15mins rest, a baseline, fasting blood sample will be taken for determination of serum insulin, total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, adiponectin and leptin, whole blood glucose and lactate, and plasma catecholamines, ghrelin, PeptideYY (PYY), glucagon-like peptide-1(GLP-1), triglycerides, and non-esterified fatty acid concentration. An expired breath sample will be collected into evacuated tubes for 13 labelled carbon dioxide (13CO2) determination, and a 20min baseline measurement of resting energy expenditure (REE) and respiratory exchange ratio (RER) will be then made using indirect calorimetry, with subjects wearing a mask, and both inspired and expired air being measured on every breath. Appetite assessment will be made by asking subjects to rate their hunger, desire to eat, fullness, and their prospective food intake, by placing a vertical mark on a 0-100mm linear scale. This visual analogue scale will be measured from left to right, with 0 indicating no experience of the variable (e.g. not hungry, unable to eat anything) and 100 indicating the most of each variable that they can imagine experiencing (e.g. intense desire to eat, or completely full). Values for these 4 variables will be combined to calculate a combined appetite score (CAS). Once baseline measurements have been completed, subjects will consume a mixed nutrient milkshake (Ensure Plus, Abbott Nutrition) at 5ml/kg body weight, which will be supplemented (at 1% of carbohydrate content) with 13-Carbon labelled (13C) Glucose. Arterialised venous blood samples will subsequently be taken every 10min for glucose and lactate assessment, and every 20min for assessment of serum insulin and incretin hormones. A measurement of REE and RER will be performed in the last 15min of every 30min period for the following 2 hours to assess fuel oxidation and metabolic rate, and an expired breath sample will be collected into evacuated tubes for 13CO2 determination at a later date. Subjective appetite will be assessed every 15minutes throughout using visual analogue scales, as described above, and at the end of the 2hr postprandial period subjects will be given an ad libitum pasta-based test meal and will be instructed to eat until they feel comfortably full. This meal will be comprised of cooked dried white pasta, commercially available tomato-based pasta sauce, olive oil and grated hard cheese, with a composition of 37% of total energy derived from fat, 48% carbohydrate, and 16% protein. The amount eaten will be recorded and related to subjective appetite ratings.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy subjects
* Body mass index < 25 kg/m2
* Height 158 - 190 cm
* Waist circumference < 94 cm
* Volunteers that are able to declare their willingness to participate in the entire study
* Willing to be assigned randomly to the three groups
* Successfully passing the psychological and medical screening
* competent to sign informed consent
* Slovenian social insurance
* English language fluency

Exclusion Criteria:

* Medication required that may interfere with the interpretation of the results
* Bone mineral density (as measured by DEXA) more than 1.5 standard deviations < t score
* Recent sub-standard nutritional status
* Family history of thrombosis or positive response in thrombosis screening procedure.

(Biochemical analysis of the following parameters: ATIII, High sensitive C-reactive protein, S-Akt., Factor V-Leiden, Prothrombin, Lupus-partial thromboplastin time, Factor II)

* History of: thyroid dysfunction, renal stones, diabetes, allergies, hypertension, hypocalcemia, uric acidaemia, lipidaemia, or hyperhomocysteinaemia
* Gastro-esophageal reflux disease or renal function disorder, Hiatus hernia
* History of medical illness
* Smoker within six months prior to the start of the study
* Abuse of drugs, medicine or alcohol
* Participation in another study up to two months before study onset
* No signed consent form before the onset of the experiment
* Blood donors in the past three months before the onset of the experiment
* Vegetarian and Vegans
* Migraines
* History of orthostatic intolerance
* History of vestibular disorders
* Claustrophobia
* metallic implants, osteosynthesis material
* Chronic back pain

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Postprandial whole blood glucose concentration | 2hrs
  a fasted sample and a sample taken every 10mins for 2hrs following eating, before and after 17days of intervention

SECONDARY OUTCOMES:
Postprandial serum insulin concentration | 2hrs
  a fasted sample and a sample taken every 20mins for 2hrs following eating, before and after 17days of intervention
Postprandial serum C-Peptide concentration | 2hrs
  a fasted sample and a sample taken every 20mins for 2hrs following eating, before and after 17days of intervention
Fasting serum leptin concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Fasting serum adiponectin concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Fasting serum total cholesterol concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Fasting serum LDL cholesterol concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Fasting serum HDL cholesterol concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Fasting plasmaTriacylglycerol concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Fasting plasma non-esterified fatty acids concentration | early morning fasted sample
  Early morning fasted sample taken before and on day 17 of intervention
Postprandial plasma peptide YY concentration | 2hrs
  a fasted sample and a sample taken every 20mins for 2hrs following eating, before and after 17days of intervention
Postprandial plasma Ghrelin concentration | 2hrs
  a fasted sample and a sample taken every 20mins for 2hrs following eating, before and after 17days of intervention
Postprandial plasma GLP-1 concentration | 2hrs
  a fasted sample and a sample taken every 20mins for 2hrs following eating, before and after 17days of intervention
Postprandial plasma catecholamine concentration | 2hrs
  a fasted sample and a sample taken every 20mins for 2hrs following eating, before and after 17days of intervention
Postprandial whole blood lactate concentration | 2hrs
  a fasted sample and a sample taken every 10mins for 2hrs following eating, before and after 17days of intervention
postprandial fuel oxidation | 2hrs
  A fasted measurement of respiratory exchange ratio and measures between 15-30, 45-60min, 75-90min and 105-120min after eating, before and on day 17 of intervention
postprandial resting energy expenditure | 2hrs
  A fasted measurement of resting energy expenditure and measures between 15-30, 45-60min, 75-90min and 105-120min after eating, before and on day 17 of intervention
postprandial subjective appetite | 2hrs
  A fasted measurement of combined appetite score (measured using visual analogue scales), followed by assessment every 30min for 2hrs after eating, before and on day 17 of intervention.
postprandial expired 13CO2 | 2hrs
  Collection of breath samples when fasted and every 30min for 2hrs after eating, before and on day 17 of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Mekjavic, PhD, Principal Investigator — Jozef Stefan Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Simpson EJ, Debevec T, Eiken O, Mekjavic I, Macdonald IA. PlanHab: the combined and separate effects of 16 days of bed rest and normobaric hypoxic confinement on circulating lipids and indices of insulin sensitivity in healthy men. J Appl Physiol (1985). 2016 Apr 15;120(8):947-55. doi: 10.1152/japplphysiol.00897.2015. Epub 2016 Jan 14. PMID 26769956
- [Result] Debevec T, Bali TC, Simpson EJ, Macdonald IA, Eiken O, Mekjavic IB. Separate and combined effects of 21-day bed rest and hypoxic confinement on body composition. Eur J Appl Physiol. 2014 Nov;114(11):2411-25. doi: 10.1007/s00421-014-2963-1. Epub 2014 Aug 5. PMID 25091855
- [Result] Debevec T, Simpson EJ, Mekjavic IB, Eiken O, Macdonald IA. Effects of prolonged hypoxia and bed rest on appetite and appetite-related hormones. Appetite. 2016 Dec 1;107:28-37. doi: 10.1016/j.appet.2016.07.005. Epub 2016 Jul 6. PMID 27395413